CLINICAL TRIAL: NCT04508049
Title: Quantitative Magnetization Transfer MRI for Evaluation of Renal Fibrosis
Brief Title: A Study to Evaluate Renal Fibrosis Using MRI Techniques
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Lilach O Lerman, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 19-008413; R01DK122734 (NIH)
Record Dates: First submitted 2020-08-06; First posted 2020-08-11 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Hypertension; Renovascular
MeSH Terms: conditions — Hypertension | interventions — Tomography, X-Ray Computed

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Early identification of fibrosis. (Other): A pilot study to test the ability of qMT to quantify fibrosis in the post-stenotic human kidney, in comparison to innovative biomarkers of renal dysfunction and tissue damage. We will pursue the Specific Aim that qMT in stenotic human kidneys is feasible and reproducible.
  Interventions: Device: qMT-MRI to detect fibrosis.

INTERVENTIONS:
Device: qMT-MRI to detect fibrosis. — The hypothesis underlying this proposal is that qMT would reliably detect development of renal fibrosis at both 1.5T and 3.0T in subjects with RVD. Patients will be studied with MRI (for fibrosis) and CT (for renal function).
  Other Names: CT scanning

SUMMARY:
The purpose of this study is to evaluate whether or not an MRI technique (quantitative magnetization transfer or qMT) in narrowing human kidneys is feasible, reproducible, and predicts recovery.

DETAILED DESCRIPTION:
Renal fibrosis is a final pathway and important biomarker of injury common to most forms of kidney disease. For example, in renal vascular disease (RVD) progressive renal fibrosis may induce kidney injury and hypertension. Early identification of fibrosis and adequate intervention may slow down renal disease progression, but adequate noninvasive strategies to detect and quantify renal fibrosis are yet to be identified.

Magnetization transfer imaging (MTI) magnetic resonance imaging (MRI) is a novel noninvasive method to evaluate the tissue macromolecular composition. The investigators have demonstrated that MTI can assess stenotic kidney fibrosis in murine and swine models of unilateral RVD. However, the clinical utility of MT-MRI to assess renal fibrosis is currently limited, because it is inherently semi-quantitative. In contrast, quantitative MT (qMT), based on biophysical compartment models, provides more objective measurement of tissue MT properties. A model fitting of MR signal acquired with various MT pulse amplitudes and offset frequencies, combined with scan-specific B0/B1/T1 maps, give rise to a more complete definition of tissue parameters, including a "bound pool fraction", a direct measure of the macromolecular content in tissue.

The hypothesis underlying this proposal is that qMT would reliably detect development of renal fibrosis at both 1.5 T and 3.0 T in subjects with RVD. To test this hypothesis, which is supported by strong preliminary data, the investigators will initially develop, optimize, and validate qMT for evaluation of fibrosis in the post-stenotic swine kidney. The investigators will correlate qMT-derived renal fibrosis with reference standards, as well as with single-kidney hemodynamics, function, and oxygenation, quantified using cutting-edge multi-detector CT (MDCT) and MRI techniques. The investigators will then determine the ability of qMT to predict renal recovery in pigs with RVD undergoing revascularization. Further, they will perform a pilot study to test the ability of qMT to quantify fibrosis in the post-stenotic human kidney, in comparison to innovative biomarkers of renal dysfunction and tissue damage.

Three specific aims will test the hypotheses: Specific Aim 1: qMT in stenotic swine kidneys is feasible, reliable, and reproducible at 1.5 and 3.0 T. Specific Aim 2: qMT predicts renal recovery potential in response to percutaneous transluminal renal angioplasty (PTRA). Specific Aim 3: qMT in stenotic human kidneys is feasible, reproducible, and predicts recovery.

The proposed studies may therefore establish a reliable, noninvasive, and clinically feasible strategy to quantify kidney fibrosis, a key biomarker for renal outcomes and therapeutic success.

ELIGIBILITY:
Inclusion Criteria:

* Between ages 40 and 80 years old.
* Patients with hypertension (BP>140/90 mmHg) and/or requirement for two or more antihypertensive medications for more than 4 weeks.
* Serum creatinine under 2.2 and 2.0 mg/dL for men and women, respectively (Caucasians). Values for African-American subjects are slightly higher (2.4 mg/dL, males; 2.1 mg/dL females).
* No contraindications to angiography: severe contrast allergy.
* No contraindications to no-contrast MR evaluations: e.g. pacemaker or magnetically active metal fragments, claustrophobia.
* Patients have the ability to comply with protocol
* Patients are competent and able to provide written informed consent

Exclusion Criteria:

* Patient has serum creatinine >2.2 mg/dL for men and >2.0 mg/dL for women (Caucasians); >2.4 mg/dL for men and >2.1 mg/dL for women (African American).
* RVD in a solitary kidney
* Patients have clinically significant medical conditions within the prior six months: e.g. myocardial infarction, congestive heart failure, stroke, that would, in the opinion of the investigators, compromise the safety of the patient.
* Uncontrolled hypertension (Systolic BP >180 mmHg despite therapy).
* Diabetes requiring insulin or oral hypoglycemic medications.
* Evidence of hepatitis B or C, or HIV infection.
* Requirement for potentially nephrotoxic drugs; e.g., non-steroidal anti-inflammatory drugs.
* Cardiac ejection fraction less than 30%.
* History of deep venous thrombosis within 3 months of enrollment.
* Kidney transplant.
* Pacemaker, implantable defibrillator or other contraindication to MRI
* Inability to comply with breath-hold for 20 seconds
* Any active malignancy and undergoing therapy
* Patients are pregnant.
* Kidney or ureteric stone
* Another known acute or chronic kidney disease
* Federal medical center inmates.
* Latex allergy

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Fibrosis assessed by qMT-MRI in the stenotic kidney and contralateral kidneys | Baseline
  A significant difference in qMT bound pool fraction (f, %) in the stenotic compared to the contralateral kidney in RVD patients.

SECONDARY OUTCOMES:
Fibrosis assessed by qMT-MRI compared to stenotic kidney function | Baseline
  A significant correlation between qMT bound pool fraction (f, %) with function (SK-GFR) and oxygenation (SK-R2*) in the stenotic kidney.
Fibrosis assessed by qMT-MRI compared to stenotic kidney injury markers | Baseline
  A significant correlation between qMT bound pool fraction (f, %) with levels of renal injury markers: Neutrophil gelatinase-associated lipocalin (NGAL), kidney injury molecular (KIM)-1, lactate dehydrogenase (LDH)], as well as urinary levels of extracellular vehicles (EVs) (measured by flow cytometry, %) originating from renal microvessels.

CONTACTS AND LOCATIONS:
Overall Officials: Lilach O Lerman, MD, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials